CLINICAL TRIAL: NCT04661969
Title: "Outcomes of Surgical Removal of Foreign Body Granulomas Due to Polymer Injection for Cosmetic Purposes"
Brief Title: "Outcomes of Surgical Removal of Foreign Body Granulomas"
Status: Completed | Type: Observational
Sponsor: Hospital Angeles del Pedregal (Other)
Responsible Party: Principal Investigator, javier lopez, Principal investigator, Plastic and reconstructive surgeon staff, MBA, FACS, Hospital Angeles del Pedregal
Other Study IDs: Polymer removal
Record Dates: First submitted 2020-12-04; First posted 2020-12-10 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Foreign Body Granuloma; Surgery; Complication
Keywords: disease-free; autoimmune/inflammatory syndrome induced by adjuvants (ASIA); adjuvant disease
MeSH Terms: conditions — Granuloma, Foreign-Body; Arthritis, Experimental | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1: Foreign Substance disseminated to both lower extremities and buttocks
  Interventions: Procedure: Surgery
- 2: Foreign Substance isolated to buttocks with moderate to severe skin changes
  Interventions: Procedure: Surgery
- 3: Foreign substance isolated to lower legs with mild skin changes and superficial ulcerations
  Interventions: Procedure: Surgery
- 4: Foreign substance isolated to lower legs with moderate to severe skin changes and/or ulceration
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Surgery — (group 1) In-bloc excision and primary closure (group 2), Resection plus Vacuum assisted closure (VAC) and split thickness skin graft (STSG) (group 3) and In-bloc excision and microsurgical reconstruction (group 4).

SUMMARY:
Illicit subcutaneous injection of high-viscosity fluids for restoration and improvement of body contour is a growing trend all around the world. Many local and systemic complications have been described. Local complications include deformity at the site of injection, granulomas and several skin changes like erythema, induration, and plaques (well-circumscribed, elevated, superficial, solid lesion).

The investigator designed a single-center, cross-sectional, retrospective, consecutive case series study and evaluated 49 surgeries performed in 35 patients with the history of foreign substances injection for cosmetic purposes and developed local complications. Investigators divided 4 groups accordingly to localization of foreign substances (FS). Group 1) FS disseminated to both lower extremities and buttocks; group 2) FS isolated to buttocks with moderate to severe skin changes, Group 3) FS isolated to lower legs with mild skin changes and superficial ulcerations and 4) FS isolated to lower legs with moderate to severe skin changes and/or ulceration. The investigators treated all patients surgically, which consisted of isolate ultrasonic liposuction for extraction of the material from the affected region (group 1) In-bloc excision and primary closure (group 2), Resection plus Vacuum assisted closure (VAC) and split thickness skin graft (STSG) (group 3) and In-bloc excision and microsurgical reconstruction (group 4). Statistical analysis was performed to find relations between type of surgery with complications, reactivation of symptoms, time for reactivation and a disease-free survival test (kaplan meier) was done.

ELIGIBILITY:
Inclusion Criteria:

* History of injection of foreign substances for cosmetic purposes
* Develop symptoms of Autoimmune syndrome induced by adjuvants
* Mild to severe skin changes

Exclusion Criteria:

* Refuse to participate in the analysis

Ages: 24 Years to 64 Years | Sex: Female
Age Groups: Adult
Study Population: patients previously injected with foreign substances (FS) such as polymers for cosmetic soft tissue augmentation and the diagnosis of ASIA presented with mild to severe skin changes and treated surgically from January 2014 to March 2020 all in a private practice setting (Hospital Angeles Pedregal, Mexico city, MEXICO) and treated all by plastic surgeon senior author (JLM)
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Complications | 30 days
  Describe if patients have or not postoperative complications

SECONDARY OUTCOMES:
Reactivation of symptoms | 9 to 76 months
  Relapse of symptoms or new local complications
Time for reactivation of symptoms | 9 to 76 months
  Account the number of months for reactivation of symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Angeles Pedregal, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Share complications table, kaplan-meier test.